CLINICAL TRIAL: NCT03924232
Title: The Bioelectrical Impedance Analysis and Muscular Ultrasound in the Detection of Nutritional Status in Critically Ill Patients: The BUS Study
Brief Title: The BIA and MUS in the Detection of Nutritional Status in Critically Ill Patients
Acronym: BUS
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, professor, University of Milan
Other Study IDs: BUS
Record Dates: First submitted 2019-04-16; First posted 2019-04-23 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: MUSCULAR AQUIRED WEAKNESS; Bioelectrical Impedance Analysis; Muscular Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Critically ill patients are characterized by wide variations in their carbohydrate, lipid, and protein metabolism. Such variations can lead to increase in their energy requirement with accelerated protein catabolism and ultimately alterations of their immune and gastrointestinal systems, and in a variable frame time, it lead to a disruption of muscular function that increased the ICU and hospital stay and mortality. There are multiple methods to conduct these measurements. However, the accuracy of these measures could be very scares. Skeletal muscle wasting in the critically ill is often masked by fluid retention. For these reasons, in the last few decades, several different tools have been developed to integrate the clinical and biochemical nutritional evaluations. Among these, the bioimpedance analysis (BIA) and the muscular ultrasonography (MU) seem to be promising tools for this purpose.

The aim of this project is to compare and integrate the data collected by BIA and MU and the routinely clinical used parameters of nutrition to define the nutritional status of critically ill patients. The data from these tools and the biochemical and anthropometric nutritional data (including the nutritional support) will be collected at the admission in ICU and followed up within the first week of ICU stay.

DETAILED DESCRIPTION:
the Bioelectrical impedance analysis and muscular Ultrasound in the detection of nutritional Status in critically ill patients

Critically ill patients are characterized by wide variations in their carbohydrate, lipid, and protein metabolism. Such variations can lead to increase in their energy requirement with accelerated protein catabolism and ultimately alterations of their immune and gastrointestinal systems, and in a variable frame time, it lead to a disruption of muscular function that increased the ICU and hospital stay and mortality. It has been observed that most of the critically ill patients who survive acute respiratory distress syndrome have to deal with a wide variety of consequences, including muscular wasting and weakness, and these conditions could last for at least one year. Intensive care unit acquired weakness has been defined as generalized weakness that develops during critical illness and where no other explanation than critical illness is present and is associated with long-term consequences from the medical, human, and socioeconomic point of view. In the normal weight person, the metabolic response to injury causes an increase in protein and energy requirements. As a result, endogenous substrates serve as fuel sources and as precursors for protein synthesis. From the nutrition perspective, one of the main challenges of providing nutritional support to critically ill patients is to stop or slow lean mass losses. For these reasons, it is fundamental for the nutritional support clinician to be able to measure and assess muscle wasting during critical illness, using an easy and accessible technique.

There are multiple methods to conduct these measurements. Usually, admission weight and height should be used to calculate the ideal body weight (IBW), the percentage of IBW, and the Body Mass Index (BMI). However, the accuracy of these measures could be very scares. Skeletal muscle wasting in the critically ill is often masked by fluid retention. In these circumstances the normal anthropometric methods of assessing changes in body mass and composition are not applicable, as the techniques all assume a normal state of hydration. Thus, additional anthropometric data although useful in ambulatory patients, are not as accurate measures of malnutrition in the critically ill patients. Moreover, some serum proteins (such as albumin level and several other transport proteins) are commonly measured as surrogates of visceral protein status. However, all of them are influenced by many factors such as synthesis and degradation rates and vascular losses into the surrounding interstitium, in addition to losses through the gut or kidney. As a result, their levels drop by inflammation or sepsis where high levels of interleukin-6 stimulate acute phase protein production as it inhibits transport protein production. Thus, they are a poor indicator of critically ill patients' nutritional status as they serve as a marker of injury and metabolic response to stress. For these reasons, in the last few decades, several different tools have been developed to integrate the clinical and biochemical nutritional evaluations. Among these, the bioimpedance analysis (BIA) and the muscular ultrasonography (MU) seem to be promising tools for this purpose.

The aim of this project is to compare and integrate the data collected by BIA and MU and the routinely clinical used parameters of nutrition to define the nutritional status of critically ill patients. The data from these tools and the biochemical and anthropometric nutritional data (including the nutritional support) will be collected at the admission in ICU and followed up within the first week of ICU stay.

Bioimpedance analysis

Bioelectrical impedance analysis (BIA) is the collective term that describes the non-invasive methods to measure the electrical body responses to the introduction of a low-level, alternating current. Recently, advances in BIA technology gave rise to detailed and sophisticated data analyses and targeted applications in clinical practice included the critical care environment. The Bioelectric Impedance Vector Analysis (BIVA) is today a commonly used approach for body composition measurements and assessment of clinical condition and has recently been developed to assess both nutritional status and tissue hydration.

Basically, BIA measures the opposition of body tissues to the flow of a small alternating current (i.e. the impedance). The classical BIA method consists of the use of four electrodes attached to the hands, wrist, foots and ankles in which a painless electrical current at a fixed or multiple frequency is introduced in the organism. Thus, BIA only measures the end to-end voltage across the entire path between the voltage-sensing electrodes. This voltage is the energy expended per unit of charge for the total current path and it does not provide any direct information with respect to the amount of current traveling through intracellular versus extracellular volumes, in blood versus muscle, or in fat versus fat-free media. The impedance is a function of two components (or vectors): the "resistance" (R) of the tissues themselves and the additional opposition or "reactance" (Xc).

Bioimpedance in the Nutritional assessment The metabolic response to critical illness is characterized by increased energy expenditure, proteolysis, gluconeogenesis and myolysis with an increment that exceeds 100% of predicted energy expenditure. This prediction can be influenced by volume overload, since body weight is often used in equations to predict energy needs. Increased proteolysis leads to accelerated protein loss, which occurs despite provision of exogenous protein and non-protein intakes. Thus, muscle wasting often occurs due to increased metabolic demands on the body, determining major losses of lean tissue due to severity of illness and organ dysfunction, prolonged immobility, and malnutrition. The variability of BIA measurements has often been cited as a major limitation for its clinical use in evaluating nutritional status. Moreover, the oldest studies were performed using a classical BIA to determine the body composition while the more recent studies focused the attention on the use of BIVA and phase angle (PA) analysis.

Bedside muscular ultrasonography in critically ill patients With growing interest in understanding muscle atrophy and function in critically ill patients and survivors, ultrasound is emerging as a potentially powerful tool for skeletal muscle quantification. It represents a simple, non-invasive method of quantification not only of central muscular (such as the diaphragm) contractile activity, but also for the peripheral skeletal muscle atrophy. This muscle quantification combined with metabolic, nutritional, and functional markers will allow optimal patient assessment and prognosis. It is now well accepted how to assess the diaphragm excursion and diaphragm thickening during breathing and the meaning of these measurements under spontaneous or mechanical ventilation, as well as features of skeletal muscle (including muscle quantity measures like mass and cross-sectional area and muscle quality measures such as architecture and evidence of myonecrosis) may provide a more feasible and objective approach to assessing muscle health in ICU patients. Moreover, objective quantifications of muscle (which include, but are not limited to, muscle mass, thickness, and cross-sectional area) that are sufficiently sensitive to detect small changes over acute timeframes may ultimately facilitate evaluation of interventions to counter muscle atrophy and weakness.

The diaphragmatic evaluation The relative contribution of patient effort during assisted breathing is difficult to measure in clinical conditions. Moreover, the diaphragm is inaccessible to direct clinical assessment. Bedside ultrasonography, which is already crucial in several aspects of critically illness has recently been proposed as a simple, non-invasive method of quantification of diaphragm contractile activity. Ultrasound can be used to determine diaphragm excursion, which may help to identify patients with diaphragm dysfunction.

Ultrasonographic examination can also allow for the direct visualization of diaphragm thickness in its zone of apposition. Thickening during active breathing has been proposed to reflect the magnitude of diaphragm effort, similarly to an ejection fraction of the heart.

A number of recent studies employed ultrasound to measure diaphragm thickness and inspiratory thickening in ventilated patients. Some of them focused on the feasibility and reproducibility of the technique, while other36 showed how with increasing levels of pressure support (PSV), parallel reductions were found between diaphragm thickening and both diaphragm and esophageal pressure-time product suggesting that diaphragm thickening is a reliable indicator of respiratory effort.

Measurement of diaphragm thickness The right hemidiaphragm can be visualized in the zone of apposition of the diaphragm to the rib cage with the probe placed in the midaxillary line, between the 8th and 10th intercostal space, as a 3-layered structure consisting of pleural and peritoneal (hyperechogenic) membranes and the hypoechogenic layer of muscle itself. This site is ideal for ultrasonographic visualization, since the diaphragm is bounded by soft tissue on either side and lies parallel to the skin surface and, therefore, the transducer face. The diaphragm is additionally dynamically identified as the most superficial structure that is obliterated by the leading edge of the lung upon inspiration. Eventually, it is identified by direct visualization of its contraction at the beginning of the respiratory cycle.

B-mode Using a 7.5-10 MHz linear probe, set in B-mode and placed parallel to a intercostal space between the VIII and X, the inferior edge of costophrenic angle is identified by the transient appearance of the lung artifact with breathing. Diaphragm thickness (Tdi) can be measured both during tidal breathing and during a maximal inspiratory effort. Several studies were performed to establish reference values of Tdi in supine healthy subjects, showing for the right hemidiaphragm mean values of 0.3238 cm or 0.3339 cm, independently of sex, age or body constitution.

M-mode The probe is placed with the same landmark previously described for B-mode with the aim to identify pleural and peritoneal membranes around the diaphragm. Diaphragm thickness is measured at end-expiration (Tdi,ee) and peak inspiration (Tdi,pi) as the distance between the diaphragmatic pleura and the peritoneum using M-mode .

Peripheral muscular assessment It has been shown that muscle mass measurement by ultrasonography (US) is a reliable technique in most of the patients even when oedema and fluid retention are present. Muscle mass loss in critically ill patients has been assessed by US, histological, and molecular biology techniques, showing a significant reduction of approximately 10% of the rectus femoris (RF) cross-sectional area (CSA) measured by US correlating with a decrease in muscle fibres CSA and less protein synthesis. US has become a widely used research technique to quantify muscle wasting showing remarkable accuracy and reliability with strong clinimetric properties and excellent intra- and interobserver reliability in healthy people measured by clinicians with no previous experience in US45.

The lower limbs muscles are prone to early atrophy, showed by a greater decrease of thickness within the first five days of admission to the intensive care unit compared with upper limbs, making these muscles a good target for muscle mass assessment.

The quadriceps femoris is a group of muscles composed by three vastus muscles (medialis, intermedius, and lateralis) and the RF. The latter one presents a proximal insertion in the anterior inferior iliac spine (AIIS) and other insertion in the supra-acetabular sulcus. The quadriceps femoris is distally inserted in the tibial tuberosity by a common ligament and is a hip flexor and a knee extensor. Before starting, make sure the patient is in supine position with extended knees and toes pointing to the ceiling. This is the most used position in this kind of measurements. This position helps the practitioner to place the patient in the AIIS Patella 1/2 AIIS Patella 1/2 1/3 1/3.

A specific technique technique has been proposed: using a non-stretchable measuring tape, trace an imaginary line in the anterior part of the thigh from the AIIS to the midpoint of the proximal border of the patella and mark the middle and one third point between these two references which easily give us access to the RF and VI. The reason to use de AIIS and not the anterior superior iliac spine is because using the exact middle point of the muscle helps us to find its thickest part using as reference the insertion points of this muscle (RF) and the reason to use a third of the distance will be discussed latter. To obtain a cross-sectional image, the transducer must be oriented transversally to the longitudinal axis (the imaginary line marked before) of the thigh forming a 90∘ angle in relation to the skin surface. Tilting or moving the probe from its original position and angle will contribute to obtaining an incorrect measurement.

Methodology The aim of the present study is to investigate and compare the diaphragmatic thickness and the cross sectional area of the rectus assessed with ultrasound using the above mentioned methodology and the data collected from BIVA as well as the nutritional and anthropometrics parameters routinely used in clinical practice. The investigators will study consecutive mechanically ventilated patients admitted in the ICU of our teaching hospital. The investigators will screen each consecutive patient who required mechanical ventilation for at least 72 hours. Non-inclusion criteria will be age <18 years, pregnancy, prevision of ICU stays less than 7 days, history/diagnosis of neuromuscular disease. Within the first 24 hours of ICU admission (T1), patients will be evaluated with muscular ultrasonography comprehensive of diaphragm thickness and rectus femoris (medial vastus) cross-sectional area. At the same time, anthropometric measure will be collected (such as body height, ideal body weight, real body weight declared, right arm circumference) as well as BIVA measure (Xc, R, PA, lean body weight and % of extracellular body weight) and biochemical analysis (inclusive albumin, pre-albumin, blood count, lymphocyte count, magnesium, phosphorus, reticulocytes, renal and hepatic function test). The day after, the fluid balance will be calculated as well as the nitrogen balance. All the same measures will be repeated at day 3 (T3) and 7 days (T7).

The main outcome of the study is to evaluate the derived BIVA parameters, especially the variation of PA, within the first week after ICU admission. The secondary outcomes are to evaluate the BIVA parameters variations and the "central" and "peripheral" muscular sonographic parameters as well as the anthropometric and biochemical nutritional indexes and their eventually correlations.

Statistical Analysis

Data will be analyzed using Stata/SE 12.0 (StataCorp, College Station) statistical software package. Normality will be assessed by the Shapiro-Francia test. Results will be reported as mean¬ ± standard deviation if normally distributed, or median [25-75th percentiles] otherwise. Comparison between related variables will be performed by paired Student's t-test or Wilcoxon sign-rank test, as needed. Two-tailed p values less than 0.05 will be considered statistically significant. The computation of the study power is based on the primary outcome. In a previous study, Kim and colleagues49 evaluated the variation of the PA in critically illness patients and the mean PA value was 3.5±1.5. Assuming a variation of 20% of the PA within the first week, a total sample size of 97 patients is calculated for 80% power at a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 or older and with a recent (<48h) ICU entry requiring mechanical ventilation for at least 3 days will be considered for enrolment

Exclusion Criteria:

* not intubated patients
* patients with an ICU prevision of stay less than 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
phase angle (PA) | one week
  variations of phase angle detected by BIVA and comparison within one week of ICU stay

SECONDARY OUTCOMES:
peripheral muscular ultrasound | one week
  Cross sectional area (CAS) of rectus femoris
Diaphragm ultrasound | one week
  Thikness Ratio (TR) of the diaphragm within one week of ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Paolo - Polo Universitario, ASST Santi Paolo e Carlo, Milan, MI, Italy